CLINICAL TRIAL: NCT05905250
Title: An mHealth Positive Psychology Intervention to Reduce Cancer Burden in Young Adult Cancer Survivors
Brief Title: mHealth for Young Adult Cancer Survivors
Acronym: mHealthAYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carla Berg, Professor of Prevention and Community Health, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCR224269; R21CA261884 (NIH)
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Survivorship; Cancer; Psychological Well-Being
MeSH Terms: conditions — Neoplasms; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Individual randomized control trial with 1:1 randomization
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigative team will be masked except in the event interventionists or data collectors require input from the team that requires disclosure of identifying information. Participants will be randomized to the intervention or attention control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention utilizes an empirically supported protocol, further refined with evidence-based strategies targeting the needs of young adult (YA) survivors. Its long-term goal is to promote hopeful thinking, and ultimately enhance other long-term markers of quality of life (QOL) (including mental health and health behaviors). The intervention follows 8 weekly curricula, reinforced through psychoeducation and skill-building, homework/practical application, and self-monitoring. Its 8-week design was informed by cognitive behavioral therapy and positive psychology intervention literature.
  Interventions: Behavioral: an empirically supported protocol, further refined with evidence-based strategies
- Attention Control (Active Comparator): Health education regarding maintaining a healthy weight, physical activity, and nutrition, based on American Cancer Society and NCI guidelines/recommendations.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: an empirically supported protocol, further refined with evidence-based strategies — The intervention utilizes an empirically supported protocol, further refined with evidence-based strategies targeting the needs of young adult (YA) survivors. Its long-term goal is to promote hopeful thinking, and ultimately enhance other long-term markers of quality of life (QOL) (including mental health and health behaviors). The intervention follows 8 weekly curricula, reinforced through psychoeducation and skill-building, homework/practical application, and self-monitoring. Its 8-week design was informed by cognitive behavioral therapy and positive psychology intervention literature.
  Arms: Intervention
Behavioral: Health education — Health education regarding maintaining a healthy weight, physical activity, and nutrition, based on American Cancer Society and NCI guidelines/recommendations.
  Arms: Attention Control

SUMMARY:
We aim to refine and pilot test an 8-week phone- and app-based intervention to promote hope, and thereby mitigate life disruption caused by cancer diagnosis and treatment, among young adults (YAs); our proposal involves (Aim 1) formative research among YA survivors and healthcare providers; and (Aim 2) an randomized controlled trial (RCT) of the intervention vs. attention control among 150 YA cancer survivors. The proposed research is innovative in its use of: 1) a novel intervention target - hope - as a mechanism for addressing goal-disruption and quality of life (QOL) among YA survivors; and 2) novel mHealth components and population-based recruitment strategy (via social media) that are particularly relevant to YA survivors and those with potentially limited access to healthcare. This proposal has potential high impact due to the number of YA cancer survivors for whom the intervention may be relevant, the intervention's potential utility in enhancing hope and QOL among YAs, and its reach/scalability.

DETAILED DESCRIPTION:
Young adulthood (YA) is a critical time in shaping life trajectories related to educational, financial, and family goals, among others. Unfortunately, cancer diagnosis/treatment and its psychosocial sequelae disrupt this critical period for some YAs. This life goal disturbance is related to poorer psychological outcomes, particularly among YAs; however, goal revision and reprioritization lead to more positive psychological outcomes. Thus, goal negotiation is a critical part of survivorship. Understanding psychosocial determinants of positive psychological and behavioral outcomes is critical for developing effective behavioral interventions. Within the rich positive psychology literature, the construct of hope is one particularly relevant factor for YA cancer survivors; hope has been defined as a positive cognitive state based on a sense of successful goal-directed determination and planning to meet these goals. In the general population and in cancer survivors, hope is related to better quality of life (QOL), mental health, health behaviors, and coping with illness/cancer. Our team pioneered an mHealth intervention (i.e., app-based with phone-based counseling) aimed at increasing hope among YA survivors, thereby re-engaging them in long-term life goals across domains (e.g., vocational, familial) and ultimately increasing QOL. In an 8-week pilot randomized controlled trial (RCT) of 56 YAs recruited from 2 cancer centers, the intervention demonstrated feasibility (95% retention), acceptability (e.g., high satisfaction), and promising trends in changes in hope, QOL, depressive symptoms, and health behaviors (e.g., substance use) in YA survivors. This study builds on our prior work to update the intervention (e.g., its technology), enhance its reach, and increase our ability to examine its effects. Our specific aims are to: 1) conduct formative research examining YA cancer survivor preferences on phone-based counseling with app support to enhance the intervention; and 2) test the feasibility, acceptability, and preliminary efficacy of the intervention vs. attention control (AC) via an 8-week RCT of 150 YA cancer survivors. The proposed research is innovative in its use of a novel intervention target - hope - as a mechanism for addressing goal-disruption and QOL among YA survivors, and its use of novel mHealth components and population-based recruitment strategy (via social media) that are particularly relevant to YA survivors and those with potentially limited access to healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I-IV cancer from age 18-39
* Completion of curative treatment (surgery, chemotherapy and/or radiation) within three years of study enrollment
* No significant psychological disabilities
* Able to complete forms and understand instructions in English
* Smartphone access
* Aim 2: Able to commit to 8-week remotely delivered study

Exclusion Criteria:

* Completion of curative treatment (surgery, chemotherapy and/or radiation) over three years ago or currently in treatment
* Significant psychological disabilities

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Berg, PhD, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Berg CJ, McCready DM, Hinds PS, Lyon ME, Dennis K, Howlader A, Bhanot P, Shajan S, Chalasani P, Chitalia A, Arem H. Outcomes of a Randomized Controlled Trial Testing the Feasibility, Acceptability and Preliminary Efficacy of a Digital, Coach-Assisted Intervention to Enhance Hope and Quality of Life Among Young Adult Cancer Survivors. Psychooncology. 2025 Nov;34(11):e70315. doi: 10.1002/pon.70315. PMID 41170949
- [Derived] Berg CJ, Schubel LC, McCready DM, Shajan S, Bhanot P, Dopke C, Howlader A, Hinds PS, Levine J, Lyon ME, Chalasani P, Arem H. Profiles of quality of life among US young adult cancer survivors and their associations with potential psychosocial intervention targets of hope and psychological flexibility. Qual Life Res. 2025 Sep;34(9):2677-2688. doi: 10.1007/s11136-025-04010-0. Epub 2025 Jun 28. PMID 40580382
- [Derived] McCready DM, Arem H, Duarte DA, Dennis K, Ball N, Cafferty LA, Hinds PS, Howlader A, Berg CJ. A digital, coach-assisted intervention to address the psychosocial needs of young adult cancer survivors: Randomized controlled trial protocol and intervention adaptation process. Contemp Clin Trials. 2024 Jun;141:107545. doi: 10.1016/j.cct.2024.107545. Epub 2024 Apr 23. PMID 38657732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study focuses on young adult (YA) cancer survivors, targeting ~150 participants total enrolled. Inclusion criteria included: 18-39 years old, within 3 years of completing primary treatment or on maintenance chemotherapy, English-speaking, US resident, and smartphone access.
Pre-assignment Details: Participants were recruited, screened for eligibility, consented, and asked to complete the baseline survey. Both AWARE and the AC involved an 8-week intervention and control for non-specific intervention components.
Period: Overall Study
Arm/Group | Intervention | Attention Control
Started | 78 | 77
Completed | 78 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Attention Control | Total
Number analyzed (Participants) | 78 | 77 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.96 (5.01) | 32.82 (4.79) | 32.89 (4.86)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at birth: female or male
  Participants
    Female | 69 | 67 | 136
    Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race, based on NIH/clinicaltrials categories
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 7 | 8 | 15
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 4 | 10
    White | 58 | 62 | 120
    More than one race | 6 | 3 | 9
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 4 | 13
  Not Hispanic or Latino | 69 | 73 | 142
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants] — US-based, recruited online
  Participants
    United States | 78 | 77 | 155
Hope [Mean (Standard Deviation); unit: units on a scale] — Hope, per Snyder's Adult Hope Scale - a 12-item measure, each scored on a 1-8 scale; 8 items assess hope-related factors (4 are distractor/filler items), for a total score range of 8-64. Higher scores indicate higher hope (better outcome).
  units on a scale | 48.74 (9.03) | 50.09 (8.03) | 49.41 (8.55)

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Number of Participants with Retention at End of Treatment
Time Frame: 2 months (end-of-treatment; EOT)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 78 | 77
Participants | 74 [70 to 78] | 72 [68 to 76]

2. Primary Outcome: Retention
Description: Number of Participants with Retention at End of Study
Time Frame: 4 months (follow-up; FU)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 78 | 77
Participants | 75 | 72

3. Primary Outcome: Adherence
Description: Adherence to intervention (number of sessions completed out of 8)
Time Frame: 2 months (end-of-treatment; EOT)
Measure: Mean (Standard Deviation); unit: Number of sessions
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 78 | 77
Number of sessions | 7.0 (2.0) [6 to 8] | 7.3 (1.8) [6 to 8]

4. Primary Outcome: Acceptability
Description: >75% participants reporting high satisfaction (3 or 4 on scale of 0=not at all to 4=very)
Time Frame: 2 months (end-of-treatment; EOT)
Population: Analyzed among participants who completed the 2-month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 74 | 72
Participants | 57 | 43

5. Primary Outcome: Acceptability
Description: >75% report yes to "would you recommend this program to your friends who are cancer survivors?"
Time Frame: 2 months (end-of-treatment; EOT)
Population: Analyzed among participants who completed the 2-month survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 74 | 72
Participants | 67 | 60

6. Primary Outcome: Hope
Description: Hope, per Snyder's Adult Hope Scale - a 12-item measure, each scored on a 1-8 scale; 8 items assess hope-related factors (4 are distractor/filler items), for a total score range of 8-64. Higher scores indicate higher hope (better outcome).
Time Frame: 4 months (follow-up; FU)
Population: Analyzed among participants who completed the 4-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 75 | 72
Scores on a scale | 50.15 (7.94) | 51.11 (8.35)

7. Secondary Outcome: Hope
Description: as for outcome 6
Time Frame: 2 months (end-of-treatment; EOT)
Population: Analyzed among participants who completed the 2-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Attention Control | Intervention
Number analyzed (Participants) | 72 | 74
Scores on a scale | 50.78 (8.32) | 49.82 (8.60)

8. Secondary Outcome: Quality of Life - Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Scale
Description: Higher scores indicate higher Quality of Life (QOL; scale 0-100) (PMCID: PMC2724630); mean scores across QOL dimensions (physical functioning, social functioning, pain interference, fatigue, sleep disturbance, anxiety, depression)
Time Frame: 2 months (end-of-treatment; EOT)
Population: Analyzed among participants who completed the 2-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 74 | 72
Scores on a scale | 51.72 (3.75) | 51.38 (3.40)

9. Secondary Outcome: Quality of Life - Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Scale
Description: Higher scores indicate higher Quality of Life (QOL; scale 0-100) (PMCID: PMC2724630); mean score across QOL dimensions (physical functioning, social functioning, pain interference, fatigue, sleep disturbance, anxiety, depression)
Time Frame: 4 months (follow-up; FU)
Population: Analyzed among participants who completed the 4-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 75 | 72
Scores on a scale | 51.17 (3.50) | 51.56 (3.10)

10. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G)
Description: Higher scores indicate higher Quality of Life (QOL; scale: 0-108) (https://www.facit.org/measures/fact-g)
Time Frame: 2 months (end-of-treatment; EOT)
Population: Analyzed among participants who completed the 2-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 74 | 72
Scores on a scale | 77.49 (17.52) | 80.17 (15.87)

11. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G)
Description: Higher scores indicate higher Quality of Life (QOL; scale: 0-108) (https://www.facit.org/measures/fact-g)
Time Frame: 4 months (follow-up; FU)
Population: Analyzed among participants who completed the 4-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 75 | 72
Scores on a scale | 79.18 (11.37) | 79.15 (10.41)

12. Secondary Outcome: Depression and Anxiety Symptoms - Mean Patient Reported Outcome Measures for Anxiety and Depression Subscales (2-month)
Description: Higher scores indicate lower anxiety and depressive symptoms (scale 0-100); mean score of across anxiety and depressive symptom subscales
Time Frame: 2 months (end-of-treatment; EOT)
Population: Analyzed among participants who completed the 2-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 74 | 72
Scores on a scale | 53.62 (8.69) | 52.68 (7.90)

13. Secondary Outcome: Depression and Anxiety Symptoms - Mean Patient Reported Outcome Measures for Anxiety and Depression Subscales (4-month)
Description: as for outcome 12
Time Frame: 4 months (follow-up; FU)
Population: Analyzed among participants who completed the 4-month survey
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention | Attention Control
Number analyzed (Participants) | 75 | 72
Scores on a scale | 52.05 (8.71) | 53.04 (8.13)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 20 weeks
Description: This study used the clinicaltrials.gov definition of adverse event and serious adverse event.
Arm/Group | Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/77
Other Adverse Events (participants affected / at risk) | 0/78 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-10-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT05905250/Prot_SAP_ICF_000.pdf